CLINICAL TRIAL: NCT02954848
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-438 10 mg Once-daily in the Treatment of Non-Erosive Gastroesophageal Reflux Disease
Brief Title: Phase 3 Study of TAK-438 10 mg in the Treatment of Non-Erosive Gastroesophageal Reflux Disease (NERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vonoprazan-3001; U1111-1188-1784 (Other: WHO); JapicCTI-163413 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease
Keywords: Drug therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): TAK-438 placebo-matching tablets, orally, once daily after breakfast for 1 week in run-in period followed by TAK-438 placebo-matching tablets, orally, once daily after breakfast for up to 4 weeks in treatment period.
  Interventions: Drug: Placebo
- TAK-438 10 mg (Experimental): TAK-438 placebo-matching tablets, orally, once daily after breakfast for 1 week in run-in period followed by TAK-438 10 mg tablets, orally, once daily after breakfast for up to 4 weeks in treatment period.
  Interventions: Drug: Placebo; Drug: TAK-438 10 mg

INTERVENTIONS:
Drug: Placebo — TAK-438 placebo-matching tablets
Drug: TAK-438 10 mg — TAK-438 tablets
  Arms: TAK-438 10 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of oral TAK-438 10 mg once-daily in the treatment of non-erosive gastroesophageal reflux disease (NERD).

DETAILED DESCRIPTION:
A phase 3, randomized, double-blind, placebo-controlled, parallel-group, multi-center study will be conducted to verify the superiority of TAK-438 (TAK-438 10 mg, once daily, 4 weeks) to placebo (placebo, once daily, 4 weeks) in participants with non-erosive gastroesophageal reflux disease (NERD).

The study consists of a 1-week, single-blind run-in period and a 4-week, double-blind treatment period. The participants will receive the study drug (TAK-438 placebo tablet) for the 1-week single-blind run-in period. After the run-in period, eligible participants will be randomized into TAK-438 10 mg or placebo treatment groups in a 1:1 ratio. The randomized participants will receive the assigned study drug (TAK-438 10 mg tablet or placebo tablet) for the 4-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written informed consent form prior to the initiation of any study procedures.
3. The participant with NERD.
4. The participant is endoscopically confirmed to have the modified Los Angeles (LA) Classification Grade N or M at the start of the run-in period (Visit 1).

   To allow efficacy evaluation in the participants with Grade N as well as in those with Grade M, the target number of participants in each grade is at least 30% of the total number of participants. Enrollment of patients with either Grade N or M will end when the number of enrolled participants with each grade exceeds 332, or 70% of the total planned number of participants.
5. The participant experiences recurrent heartburn, on at least 2 days a week over the last 3 weeks prior to the start of the run-in period (Visit 1).
6. The participant is either a male or female outpatient with a minimum age of 20 years at the time of informed consent signing. However, participants who are hospitalized only for examination purposes are also allowed to participate.
7. A female participant of childbearing potential agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study, and for 4 weeks after the last dose of study drug.
8. The participant's compliance to the study drug has been good (75% or better) in the run-in period.
9. The participant has experienced heartburn on at least 2 days in the last 1 week prior to randomization.
10. The participant has appropriately provided in the patient's diary all the required information during the run-in period.

Exclusion Criteria:

1. The participant has received any investigational compound within 84 days prior to the first dose of study drug.
2. The participant has received TAK-438 in a previous clinical study or as a therapeutic agent, except one with experience of receiving TAK-438 as an adjunct therapy for H. pylori eradication, who can be enrolled in this study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The participant has donated at least 400 mL of blood within the 90 days prior to the start of the run-in period (Visit 1).
5. Endoscopic examination for entering this study fails to diagnose NERD within 84 days before the start of the run-in period (Visit 1).
6. The participant has any complications affecting the esophagus, including Barrett's esophagus (3 cm or more, long segment Barrett's esophagus [LSBE]), eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, and esophageal stenosis; a history of radiation therapy or cryotherapy for the esophagus; or caustic or physiochemical trauma (eg, esophageal sclerotherapy). However, participants with Barrett's mucosa (less than 3 cm, short segment Barrett's esophagus [SSBE]) or Schatzki's ring (a mucosal tissue ring lining the inferior esophageal sphincter) are permitted to participate.
7. The participant has a history of surgery or treatment affecting gastroesophageal reflux, including fundoplication and mechanical dilatation for esophageal stenosis (except Schatzki's ring), or a history of gastric or duodenal surgery (except endoscopic removal of benign polyps).
8. The participant has acute upper gastrointestinal bleeding or gastric or duodenal ulcer, characterized by a defective mucosa with white coating, within 30 days prior to the start of the run-in period (Visit 1). However, participants with gastric or duodenal erosion are permitted to participate.
9. The participant has acute gastritis or acute exacerbation of chronic gastritis.
10. The participant has, or has a history of, Zollinger-Ellison syndrome or gastric acid hypersecretion disorders.
11. The participant has, or has a history of chest pain due to cardiac disease, or has chest pain suspectedly caused by cardiac disease within 1 year prior to the start of the run-in period (Visit 1).
12. The participant has any other concurrent upper gastrointestinal symptoms more severe than heartburn.
13. The participant has depression.
14. The participant has, has a history of, or is suspected of functional upper gastrointestinal disorders, such as functional dyspepsia and functional heartburn diagnosed by the Rome IV criteria.
15. The participant has a history of hypersensitivity or allergies to TAK-438 (including the formulation excipients).
16. The participant has a history or complication of drug abuse (defined as any illicit drug use) or of alcohol abuse within 1 years prior to the start of the run-in period (Visit 1).
17. The participant requires any excluded medications or treatments.
18. The female participant who is pregnant, is lactating, or is intending to become pregnant or to donate ova any time between the informed consent signing and 4 weeks after the last dose of study drug.
19. The participant has any serious neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrinological, or hematologic diseases.
20. The participant needs surgery requiring hospitalization during the course of the study, or surgery requiring hospitalization is scheduled for the participant during the course of the study.
21. The participant has a history of malignancy or is treated for malignancy within 5 years prior to the start of the run-in period (Visit 1). However, participants who have recovered completely from cutaneous basal cell carcinoma or from cervical carcinoma in situ are permitted to participate.
22. The participant has acquired immunodeficiency syndrome (AIDS) or hepatitis, is a human immunodeficiency virus (HIV) carrier, or tested positive for the hepatitis B virus surface antigen (HBsAg) or the hepatitis C virus (HCV) antibody. However, participants who tested negative for HCV antigen or HCV-RNA are permitted to participate.
23. The participant has any of the following abnormal clinical laboratory test values at the start of the run-in period (Visit 1):

    * Creatinine > 2 mg/dL.
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN).
    * Bilirubin (Total bilirubin) > ULN.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- Japan (30):
  - Abiko, Chiba
  - Yachiyo, Chiba
  - Kasuya-gun, Fukuoka
  - Kitakyushu, Fukuoka
  - Wakasugi, Fukuoka
  - Yukuhashi, Fukuoka
  - Kōriyama, Fukushima
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Suzaki, Kochi
  - Kitakatsuragi, Nara
  - Fujimi, Saitama
  - Hiki-gun, Saitama
  - Satte, Saitama
  - Ōtawara, Tochigi
  - Arakawa-ku, Tokyo
  - Nakano-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Toshima-ku, Tokyo
  - Fukuoka
  - Hiroshima
  - Kochi
  - Kumamoto
  - Nagasaki
  - Osaka
  - Ōita
  - Shizuoka
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Kinoshita Y, Sakurai Y, Takabayashi N, Kudou K, Araki T, Miyagi T, Iwakiri K, Ashida K. Efficacy and Safety of Vonoprazan in Patients With Nonerosive Gastroesophageal Reflux Disease: A Randomized, Placebo-Controlled, Phase 3 Study. Clin Transl Gastroenterol. 2019 Nov;10(11):e00101. doi: 10.14309/ctg.0000000000000101. PMID 31770139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 44 investigative sites in Japan from 15 November 2016 to 26 February 2018.
Pre-assignment Details: Participants with a diagnosis of non-erosive gastroesophageal reflux disease (NERD) were enrolled and received one tablet of placebo orally, once daily in a run-in period. After that, the participants who met all the entry criteria were randomized in 1:1 ratio to receive TAK-438 10 mg or TAK-438 placebo-matching tablets.
Period: Overall Study
Arm/Group | Placebo | TAK-438 10 mg
Started | 245 | 239
Treated | 245 | 238
Completed | 243 | 234
Not Completed | 2 | 5
Not completed — Randomized but Not Treated | 0 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Participant | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-438 10 mg | Total
Number analyzed (Participants) | 245 | 239 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (15.38) | 52.8 (14.37) | 52.3 (14.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 161 | 301
  Male | 105 | 78 | 183
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 245 | 239 | 484
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  cm
    number analyzed (Participants) | 245 | 237 | 482
    (all) | 161.7 (8.62) | 160.5 (9.29) | 161.1 (8.97)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  kg
    number analyzed (Participants) | 245 | 237 | 482
    (all) | 59.6 (12.04) | 58.7 (11.15) | 59.2 (11.61)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight (kg)/[height (m)^2] Population: Number analyzed are the participants who were evaluated for this baseline measure.
  kg/m^2
    number analyzed (Participants) | 245 | 237 | 482
    (all) | 22.67 (3.431) | 22.71 (3.375) | 22.69 (3.400)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 124 | 128 | 252
  Current Smoker | 52 | 44 | 96
  Ex-smoker | 69 | 67 | 136
Consumption of Alcohol [Count of Participants; unit: Participants]
  Drank Every Day | 59 | 46 | 105
  Drank a Couple of Days Per Week | 62 | 63 | 125
  Drank a Couple of Days Per Month | 54 | 54 | 108
  Never Drank | 70 | 76 | 146
Consumption of Caffeine [Count of Participants; unit: Participants]
  Had Caffeine Consumption | 192 | 190 | 382
  Had No Caffeine Consumption | 53 | 49 | 102
Endoscopic Findings by Principal Investigator (PI) [Count of Participants; unit: Participants] — Endoscopic findings were assessed using the modified Los Angeles (LA) classification. The modified LA classification would be graded as follows- Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks <5 mm in length; Grade B: nonconfluent mucosal breaks ≥ 5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
  Participants
    Grade N | 82 | 81 | 163
    Grade M | 163 | 158 | 321
Endoscopic Findings by Central Adjudication Committee (CAC) [Count of Participants; unit: Participants] — Endoscopic findings were assessed by CAC, and participant eligibility was confirmed based on the decision by investigator. Assessments were done using modified Los Angeles (LA) classification. The modified LA classification would be graded as follows- Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: nonconfluent mucosal breaks < 5mm in length; Grade B: non-confluent mucosal breaks ≥5 mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
  Participants
    Grade M | 168 | 157 | 325
    Grade N | 77 | 82 | 159
Barrett's Mucosa [Count of Participants; unit: Participants] — Participants with Barrett's mucosa less than 3 cm were indicated as Yes (Less than 3 cm), and participants with no Barrett's mucosa were indicated as No.
  Participants
    Yes (Less than 3 cm) | 56 | 51 | 107
    No | 189 | 188 | 377
Esophageal Hiatal Hernia [Count of Participants; unit: Participants] — Participants with esophageal hiatal hernia of 2 cm or more were indicated as Yes (2 cm or More) and with those of less than 2 cm were indicated as Yes (Less than 2 cm). Participants with no esophageal hiatal hernia were indicated as No.
  Participants
    Yes (2 cm or More) | 17 | 18 | 35
    Yes (Less than 2 cm) | 82 | 85 | 167
    No | 146 | 136 | 282
Severity of Symptoms, Heartburn [Mean (Standard Deviation); unit: score on a scale] — Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity.The mean severity of heartburn was calculated by the number of severity score in daily diaries. Population: Number analyzed are the participants who were evaluated for this baseline measure.
  score on a scale
    number analyzed (Participants) | 245 | 238 | 483
    (all) | 1.641 (0.5747) | 1.765 (0.6171) | 1.702 (0.5986)
Severity of Symptoms, Regurgitation [Mean (Standard Deviation); unit: score on a scale] — Most common acid reflux symptom of non-erosive gastroesophageal reflux disease (NERD) is heartburn, followed by regurgitation. Regurgitation symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of regurgitation in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. The mean severity of regurgitation was calculated by the number of severity score in daily diaries. Population: Number analyzed are the participants who were evaluated for this baseline measure.
  score on a scale
    number analyzed (Participants) | 245 | 238 | 483
    (all) | 1.074 (0.8398) | 1.109 (0.9092) | 1.091 (0.8739)
Use of Proton Pump Inhibitors (PPIs) Within 180 Days Prior to Informed Consent (IC) [Count of Participants; unit: Participants] — The numbers of participants with the answer to the following question were indicated: Has participants taken PPIs within 180 Days prior to IC?
  Participants
    Yes | 45 | 55 | 100
    No | 200 | 184 | 384
Use of H2-Receptor Antagonists (H2RA) Within 180 Days Prior to IC [Count of Participants; unit: Participants] — The numbers of participants with the answer to the following question were indicated: Has participants taken H2RA within 180 Days prior to IC?
  Participants
    Yes | 29 | 28 | 57
    No | 216 | 211 | 427
Use of Other Agents (Anticholinergics or Anti-gastrin Drugs) within 180 Days Prior to IC [Count of Participants; unit: Participants] — The numbers of participants with the answer to the following question were indicated: Has participants taken other agents (anticholinergics or anti-gastrin drugs) within 180 Days prior to IC?
  Participants
    Yes | 24 | 22 | 46
    No | 221 | 217 | 438
Response to Acid Suppressants [Count of Participants; unit: Participants] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  Participants
    number analyzed (Participants) | 91 | 93 | 184
    Heartburn has been Resolved | 31 | 45 | 76
    Heartburn has not been Resolved but Relieved | 52 | 43 | 95
    Heartburn has Remained Unchanged | 8 | 5 | 13
Response to Acid Suppressants [Count of Participants; unit: Participants] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  Participants
    number analyzed (Participants) | 91 | 93 | 184
    Improved | 83 | 88 | 171
    Not Improved | 8 | 5 | 13
History of H. pylori Eradication [Count of Participants; unit: Participants]
  Within the Last Year | 2 | 1 | 3
  More than One Year Before | 58 | 49 | 107
  No | 185 | 189 | 374
Serological Determination for H. pylori [Count of Participants; unit: Participants] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  Participants
    number analyzed (Participants) | 245 | 237 | 482
    Positive | 37 | 28 | 65
    Negative | 208 | 209 | 417
Gastrin [Mean (Standard Deviation); unit: pg/mL] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  pg/mL
    number analyzed (Participants) | 243 | 237 | 480
    (all) | 91.6 (53.29) | 103.1 (182.68) | 97.3 (133.83)
Ratio of Pepsinogen I to Pepsinogen II [Mean (Standard Deviation); unit: ratio] — Population: Number analyzed are the participants who were evaluated for this baseline measure.
  ratio
    number analyzed (Participants) | 243 | 237 | 480
    (all) | 7.63 (2.722) | 7.57 (2.442) | 7.60 (2.585)
Factors and Improvement: Physical Factors, Kyphosis [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with physical factors of kyphosis were indicated as Yes and those with no factors were indicated as No.
  Participants
    Yes | 4 | 8 | 12
    No | 241 | 231 | 472
Factors and Improvement: Physical Factors, Evident Obesity [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with physical factors of evident obesity were indicated as Yes and those with no factors were indicated as No.
  Participants
    Yes | 14 | 15 | 29
    No | 231 | 224 | 455
Factors and Improvement: Movement, Forward Flexion [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with movement of forward flexion were indicated as Yes and those with no movement of forward flexion were indicated as No.
  Participants
    Yes | 105 | 83 | 188
    No | 140 | 156 | 296
Factors and Improvement: Movement, Lying in Bed [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of lying in bed were indicated as Yes and those with no habits of lying in bed were indicated as No.
  Participants
    Yes | 99 | 89 | 188
    No | 146 | 150 | 296
Factors and Improvement: Movement, Other [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with movement of other which caused heartburn and improvement in living habits were indicated as Yes and those with no movement of other were indicated as No.
  Participants
    Yes | 13 | 12 | 25
    No | 232 | 227 | 459
Factors and Improvement: Diet, Fatty Foods (Fried Foods, Stodge, etc.) [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking fatty foods (fried foods, stodge, etc.) were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 165 | 156 | 321
    No | 80 | 83 | 163
Factors and Improvement: Diet, Carbohydrates (Grains, Potatoes, etc.) [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking carbohydrates (grains, potatoes, etc.) were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 115 | 90 | 205
    No | 130 | 149 | 279
Factors and Improvement: Diet, Sweet Foods (Chocolate, etc.) [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking sweet foods (chocolate, etc.) were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 87 | 78 | 165
    No | 158 | 161 | 319
Factors and Improvement: Diet, Acidic Foods (Citrus Fruits, Carb. Beverage) [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking acidic foods (citrus fruits, carb. beverage) were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 79 | 66 | 145
    No | 166 | 173 | 339
Factors and Improvement: Diet, Spices (Pepper, Curry, etc.) [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking spices (pepper, curry, etc.) were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 83 | 77 | 160
    No | 162 | 162 | 324
Factors and Improvement: Diet, Other [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of taking other foods which caused heartburn and improvement in living habits were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 5 | 13 | 18
    No | 240 | 226 | 466
Factors and Improvement: Habits, Smoking [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of smoking were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 29 | 19 | 48
    No | 216 | 220 | 436
Factors and Improvement: Habits, Caffeine Ingestion [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of caffeine ingestion were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 112 | 112 | 224
    No | 133 | 127 | 260
Factors and Improvement: Habits, Drinking Alcohol [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with habits of drinking alcohol were indicated as Yes and those with no habits were indicated as No.
  Participants
    Yes | 79 | 68 | 147
    No | 166 | 171 | 337
Factors and Improvement: Above Factors are NA or cannot be Specified [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with above factors are not applicable or cannot be specified were indicated as Yes and those with factors were indicated as No. Here, NA=Not Applicable.
  Participants
    Yes | 4 | 8 | 12
    No | 241 | 231 | 472
Factors and Improvement: Improving Lifestyle [Count of Participants; unit: Participants] — Factors were included which caused heartburn and improvement in living habits. Participants with improving their lifestyle were indicated as Yes and those without improvement were indicated as No.
  Participants
    Yes | 84 | 97 | 181
    No | 161 | 142 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Without Symptoms of Heartburn
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. Reported data was the percentage of days for each group, calculated by the number of days without heartburn divided by the number of days of treatment period.
Time Frame: Up to Week 4
Population: Full analysis set (FAS) included participants who were randomized and received at least one dose of the study drug.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of days | 61.50 [0.0 to 100.0] | 72.55 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0643, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.800, 95% CI 2-sided [0.000 to 10.600] — The point estimate of the median difference between the treatment groups was calculated using the Hodges-Lehmann estimation

2. Primary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. Cumulative rate of improvement was calculated as percentage of participants who experienced symptom improvement. Symptom improvement was defined as symptoms experienced on less than 2 days of the last 7 days. The cumulative data was collected between Day 0 and Day 24 and is reported for the following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24. Data not collected were shown as NA = Not Applicable.
Time Frame: Day 0 to Day 24
Population: FAS included participants who were randomized and received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0 | 0.0 | 0.0
  Day 1 | 14.7 | 23.1
  Day 2 | 15.9 | 24.4
  Day 3 | 16.3 | 25.2
  Day 4 | 17.6 | 26.1
  Day 5 | 18.8 | 28.2
  Day 6 | 19.2 | 30.4
  Day 7 | 20.0 | 32.5
  Day 8 | 21.2 | 32.9
  Day 9 | 23.7 | 34.2
  Day 10 | NA — Data was not collected at this time point. | 35.5
  Day 11 | 25.7 | 38.5
  Day 12 | 27.3 | 41.1
  Day 13 | 29.0 | 44.6
  Day 14 | 30.6 | 46.7
  Day 15 | 31.4 | 48.9
  Day 16 | 34.3 | 49.7
  Day 17 | 36.3 | 51.0
  Day 18 | 38.4 | 54.4
  Day 19 | 40.0 | 55.7
  Day 20 | 42.7 | 59.0
  Day 21 | 44.7 | 59.5
  Day 22 | 48.6 | 62.7
  Day 23 | 51.3 | 66.1
  Day 24 | NA — Data was not collected at this time point. | 71.3
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0003, Log Rank

3. Primary Outcome: Severity of Symptoms of Heartburn
Description: Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. The severity of heartburn was calculated by the number of severity score in daily diaries.
Time Frame: Up to Week 4
Population: FAS included participants who were randomized and received at least one dose of the study drug.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
score on a scale | 1.140 [0.00 to 2.82] | 1.070 [0.00 to 3.67]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0826, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1100, 95% CI 2-sided [-0.2400 to 0.0100]

4. Secondary Outcome: Percentage of Days Without Symptoms of Heartburn in Subgroup Stratified by Response (Improved or Not Improved) at Week 2
Description: Participants recorded the presence and severity of heartburn in a daily participant diary. Percentage of days without heartburn was calculated in each subgroup of the response (improved or not improved) according to Criteria 1, i.e. Improved: the participants experienced heartburn on less than 2 days of the 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: the participants experienced heartburn on 2 days or more of the 7 days prior to Week 2 [Day 8 through Day 14] and Criteria 2, i.e. Improved: the proportion of days the participants experienced heartburn during the treatment period up to Week 2 [Day 14] was lower than that during the run-in period; Not improved: the proportion of days the participants experienced heartburn during the treatment period up to Week 2 [Day 14] was equal to or larger than that during the run-in period.
Time Frame: Up to Week 4
Population: FAS included participants who were randomized and received at least one dose of the study drug. Number analyzed is the number of participants who were evaluable at each category.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of days
  Criteria 1, Improved: number analyzed (Participants) | 83 | 99
  Criteria 1, Improved | 92.00 [41.4 to 100.0] | 96.00 [46.4 to 100.0]
  Criteria 1, Not Improved: number analyzed (Participants) | 162 | 136
  Criteria 1, Not Improved | 50.95 [0.0 to 92.9] | 48.05 [0.0 to 92.9]
  Criteria 2, Improved: number analyzed (Participants) | 168 | 174
  Criteria 2, Improved | 71.40 [3.3 to 100.0] | 81.15 [14.3 to 100.0]
  Criteria 2, Not Improved: number analyzed (Participants) | 77 | 64
  Criteria 2, Not Improved | 39.30 [0.0 to 83.3] | 24.15 [0.0 to 84.0]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 1, improved response; Test type: Superiority; p = 0.0478, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.300, 95% CI 2-sided [0.000 to 5.300]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 1, not improved response; Test type: Superiority; p = 0.8963, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.000, 95% CI 2-sided [-6.100 to 6.000]
Statistical Analysis 3: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 2, improved response; Test type: Superiority; p = 0.0120, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 5.200, 95% CI 2-sided [0.000 to 10.700]
Statistical Analysis 4: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 2, not improved response; Test type: Superiority; p = 0.0871, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -4.700, 95% CI 2-sided [-17.400 to 0.000]

5. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Improved Per Criteria 1) at Week 2
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. Cumulative rate of improvement was calculated as percentage of participants who experienced symptom improvement. The response was evaluated per Criteria 1, i.e. Improved: the participants experienced heartburn on less than 2 days of the 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: the participants experienced heartburn on 2 days or more of the 7 days prior to Week 2 [Day 8 through Day 14]. Cumulative data was collected between Day 0 and Day 22 and is reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 11, 15, 16, 17, 18, 19, 20, 21, and 22. Data not collected were shown as NA = Not Applicable.
Time Frame: Day 0 to Day 22
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 83 | 99
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 83 | 99
  Day 1 | 43.4 | 55.6
  Day 2: number analyzed (Participants) | 83 | 99
  Day 2 | 47.0 | 58.6
  Day 3: number analyzed (Participants) | 83 | 99
  Day 3 | 48.2 | 60.6
  Day 4: number analyzed (Participants) | 83 | 99
  Day 4 | 51.8 | 62.6
  Day 5: number analyzed (Participants) | 83 | 99
  Day 5 | 55.4 | 67.7
  Day 6: number analyzed (Participants) | 83 | 99
  Day 6 | 56.6 | 72.7
  Day 7: number analyzed (Participants) | 83 | 99
  Day 7 | 59.0 | 77.8
  Day 8: number analyzed (Participants) | 83 | 99
  Day 8 | 62.7 | 78.8
  Day 11: number analyzed (Participants) | 83 | 99
  Day 11 | NA — Data was not collected at this time point. | 80.8
  Day 15: number analyzed (Participants) | 83 | 99
  Day 15 | NA — Data was not collected at this time point. | 81.8
  Day 16: number analyzed (Participants) | 83 | 99
  Day 16 | 63.9 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 83 | 99
  Day 17 | 65.1 | NA — Data was not collected at this time point.
  Day 18: number analyzed (Participants) | 83 | 99
  Day 18 | NA — Data was not collected at this time point. | 83.8
  Day 19: number analyzed (Participants) | 83 | 99
  Day 19 | 66.3 | NA — Data was not collected at this time point.
  Day 20: number analyzed (Participants) | 83 | 99
  Day 20 | 69.2 | 87.6
  Day 21: number analyzed (Participants) | 83 | 99
  Day 21 | 70.6 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 83 | 99
  Day 22 | 75.5 | 93.8
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0025, Log Rank

6. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Not Improved Per Criteria 1) at Week 2
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. Cumulative rate of improvement is calculated as percentage of participants who experienced symptom improvement. The response was evaluated per Criteria 1, i.e. Improved: the participants experienced heartburn on less than 2 days of the 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: the participants experienced heartburn on 2 days or more of the 7 days prior to Week 2 [Day 8 through Day 14]. Cumulative data was collected between Day 0 and Day 24 and is reported for following time points: Days 0, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24. Data not collected were shown as NA = Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 162 | 136
  Day 0 | 0.0 | 0.0
  Day 9: number analyzed (Participants) | 162 | 136
  Day 9 | 3.7 | 2.2
  Day 10: number analyzed (Participants) | 162 | 136
  Day 10 | NA — Data was not collected at this time point. | 4.4
  Day 11: number analyzed (Participants) | 162 | 136
  Day 11 | 6.8 | 8.1
  Day 12: number analyzed (Participants) | 162 | 136
  Day 12 | 9.3 | 12.6
  Day 13: number analyzed (Participants) | 162 | 136
  Day 13 | 11.7 | 18.5
  Day 14: number analyzed (Participants) | 162 | 136
  Day 14 | 14.2 | 22.2
  Day 15: number analyzed (Participants) | 162 | 136
  Day 15 | 15.4 | 25.2
  Day 16: number analyzed (Participants) | 162 | 136
  Day 16 | 19.1 | 26.7
  Day 17: number analyzed (Participants) | 162 | 136
  Day 17 | 21.6 | 28.9
  Day 18: number analyzed (Participants) | 162 | 136
  Day 18 | 24.7 | 33.3
  Day 19: number analyzed (Participants) | 162 | 136
  Day 19 | 26.6 | 35.6
  Day 20: number analyzed (Participants) | 162 | 136
  Day 20 | 29.2 | 38.7
  Day 21: number analyzed (Participants) | 162 | 136
  Day 21 | 31.5 | 39.5
  Day 22: number analyzed (Participants) | 162 | 136
  Day 22 | 34.9 | 41.7
  Day 23: number analyzed (Participants) | 162 | 136
  Day 23 | 39.2 | 47.0
  Day 24: number analyzed (Participants) | 162 | 136
  Day 24 | NA — Data was not collected at this time point. | 55.1
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.1059, Log Rank

7. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Improved Per Criteria 2) at Week 2
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in daily participant diary. The score range was 0-4, with higher scores reflecting the greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response evaluated per Criteria 2, i.e. Improved: proportion of days participant experienced heartburn during treatment period up to Week 2 [Day 14] was lower than that during run-in period; Not improved: proportion of days participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal to or larger than that during the run-in period. Cumulative data was collected between Day 0 and Day 24 and is reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 168 | 174
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 168 | 174
  Day 1 | 21.4 | 31.6
  Day 2: number analyzed (Participants) | 168 | 174
  Day 2 | 23.2 | 33.3
  Day 3: number analyzed (Participants) | 168 | 174
  Day 3 | 23.8 | 34.5
  Day 4: number analyzed (Participants) | 168 | 174
  Day 4 | 25.6 | 35.6
  Day 5: number analyzed (Participants) | 168 | 174
  Day 5 | 26.2 | 38.5
  Day 6: number analyzed (Participants) | 168 | 174
  Day 6 | 26.8 | 41.4
  Day 7: number analyzed (Participants) | 168 | 174
  Day 7 | 28.0 | 44.3
  Day 8: number analyzed (Participants) | 168 | 174
  Day 8 | 29.8 | 44.9
  Day 9: number analyzed (Participants) | 168 | 174
  Day 9 | 32.1 | 46.0
  Day 10: number analyzed (Participants) | 168 | 174
  Day 10 | NA — Data was not collected at this time point. | 47.8
  Day 11: number analyzed (Participants) | 168 | 174
  Day 11 | 34.5 | 51.8
  Day 12: number analyzed (Participants) | 168 | 174
  Day 12 | 36.9 | 54.1
  Day 13: number analyzed (Participants) | 168 | 174
  Day 13 | 38.7 | 57.6
  Day 14: number analyzed (Participants) | 168 | 174
  Day 14 | NA — Data was not collected at this time point. | 58.2
  Day 15: number analyzed (Participants) | 168 | 174
  Day 15 | 39.3 | 60.0
  Day 16: number analyzed (Participants) | 168 | 174
  Day 16 | 42.3 | 61.1
  Day 17: number analyzed (Participants) | 168 | 174
  Day 17 | 45.3 | 62.3
  Day 18: number analyzed (Participants) | 168 | 174
  Day 18 | 47.1 | 65.2
  Day 19: number analyzed (Participants) | 168 | 174
  Day 19 | 48.3 | 66.3
  Day 20: number analyzed (Participants) | 168 | 174
  Day 20 | 50.9 | 69.5
  Day 21: number analyzed (Participants) | 168 | 174
  Day 21 | 52.4 | 70.1
  Day 22: number analyzed (Participants) | 168 | 174
  Day 22 | 56.7 | 71.9
  Day 23: number analyzed (Participants) | 168 | 174
  Day 23 | NA — Data was not collected at this time point. | 74.5
  Day 24: number analyzed (Participants) | 168 | 174
  Day 24 | NA — Data was not collected at this time point. | 78.7
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0004, Log Rank

8. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Not Improved Per Criteria 2) at Week 2
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in daily participant diary. The score range was 0-4, with higher scores reflecting the greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. The response evaluated per Criteria 2, i.e. Improved: proportion of days participant experienced heartburn during treatment period up to Week 2 [Day 14] was lower than that during run-in period; Not improved: proportion of days participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal to or larger than that during run-in period. Cumulative data was collected between Day 0 and Day 24 and is reported for following time points: Days 0, 5, 9, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 77 | 64
  Day 0 | 0.0 | 0.0
  Day 5: number analyzed (Participants) | 77 | 64
  Day 5 | 2.6 | NA — Data was not collected at this time point.
  Day 9: number analyzed (Participants) | 77 | 64
  Day 9 | 5.2 | 1.6
  Day 11: number analyzed (Participants) | 77 | 64
  Day 11 | 6.5 | NA — Data was not collected at this time point.
  Day 12: number analyzed (Participants) | 77 | 64
  Day 12 | NA — Data was not collected at this time point. | 4.9
  Day 13: number analyzed (Participants) | 77 | 64
  Day 13 | 7.8 | 8.2
  Day 14: number analyzed (Participants) | 77 | 64
  Day 14 | 13.0 | 14.8
  Day 15: number analyzed (Participants) | 77 | 64
  Day 15 | 14.3 | 18.0
  Day 16: number analyzed (Participants) | 77 | 64
  Day 16 | 16.9 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 77 | 64
  Day 17 | NA — Data was not collected at this time point. | 19.7
  Day 18: number analyzed (Participants) | 77 | 64
  Day 18 | 19.5 | 24.6
  Day 19: number analyzed (Participants) | 77 | 64
  Day 19 | 22.1 | 26.2
  Day 20: number analyzed (Participants) | 77 | 64
  Day 20 | 24.9 | 29.7
  Day 21: number analyzed (Participants) | 77 | 64
  Day 21 | 27.9 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 77 | 64
  Day 22 | 31.3 | 37.0
  Day 23: number analyzed (Participants) | 77 | 64
  Day 23 | 41.1 | 42.7
  Day 24: number analyzed (Participants) | 77 | 64
  Day 24 | NA — Data was not collected at this time point. | 50.9
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.5393, Log Rank

9. Secondary Outcome: Severity of Symptoms of Heartburn in Subgroup Stratified by Response (Improved or Not Improved) at Week 2
Description: Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, the higher scores indicates greater severity. The severity was calculated in each subgroup of response (improved or not improved) according to Criteria 1, i.e. Improved: participants experienced heartburn on less than 2 days of the 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: participants experienced heartburn on 2 days or more of the 7 days prior to Week 2 [Day 8 through Day 14] and Criteria 2, i.e. Improved: proportion of days the participants experienced heartburn during the treatment period up to Week 2 [Day 14] was lower than that during the run-in period; Not improved: proportion of days the participants experienced heartburn during the treatment period up to Week 2 [Day 14] was equal to or larger than that during the run-in period.
Time Frame: Up to Week 4
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
score on a scale
  Criteria 1, Improved: number analyzed (Participants) | 83 | 99
  Criteria 1, Improved | 0.420 [0.00 to 1.44] | 0.310 [0.00 to 1.56]
  Criteria 1, Not Improved: number analyzed (Participants) | 162 | 136
  Criteria 1, Not Improved | 1.430 [0.25 to 2.82] | 1.420 [0.14 to 2.64]
  Criteria 2, Improved: number analyzed (Participants) | 168 | 174
  Criteria 2, Improved | 0.960 [0.00 to 2.14] | 0.675 [0.00 to 2.04]
  Criteria 2, Not Improved: number analyzed (Participants) | 77 | 64
  Criteria 2, Not Improved | 1.610 [0.44 to 2.82] | 1.740 [0.43 to 3.67]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 1, improved response; Test type: Superiority; p = 0.0505, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1000, 95% CI 2-sided [-0.2100 to 0.0000]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 1, not improved response; Test type: Superiority; p = 0.8138, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.0200, 95% CI 2-sided [-0.1200 to 0.1500]
Statistical Analysis 3: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 2, improved response; Test type: Superiority; p = 0.0129, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1500, 95% CI 2-sided [-0.2800 to -0.0300]
Statistical Analysis 4: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for criteria 2, not improved response; Test type: Superiority; p = 0.0765, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.1700, 95% CI 2-sided [-0.0100 to 0.3600]

10. Secondary Outcome: Percentage of Days Without Symptoms of Heartburn in Subgroup Stratified by Endoscopic Findings (the Modified LA Classification Grade N or M) at Baseline
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, higher scores indicates greater severity. The percentage was calculated in each subgroup of the endoscopic findings where Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks <5mm in length; Grade B: non-confluent mucosal breaks ≥5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
Time Frame: Up to Week 4
Population: FAS included participants who were randomized and received at least one dose of the study drug. Number analyzed is the number of participants who had endoscopic findings.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of days
  Grade N: number analyzed (Participants) | 82 | 81
  Grade N | 64.15 [0.0 to 100.0] | 76.70 [0.0 to 100.0]
  Grade M: number analyzed (Participants) | 163 | 157
  Grade M | 60.70 [0.0 to 100.0] | 67.90 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Grade N of endoscopic findings; Test type: Superiority; p = 0.1490, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 6.500, 95% CI 2-sided [-1.900 to 15.300]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Grade M of endoscopic findings; Test type: Superiority; p = 0.2146, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.600, 95% CI 2-sided [-1.400 to 10.700]

11. Secondary Outcome: Cumulative Rate of Improvement in Heartburn in Subgroup Stratified by Endoscopic Findings (the Modified LA Classification Grade N) at Baseline
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. The score range was 0-4, higher scores indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Cumulative rate calculated in subgroup of Grade N per modified LA classification. Modified LA classification Grade N: normal mucosa; Grade M: minimal changes to mucosa; Grade A: nonconfluent mucosal breaks <5mm in length; Grade B: non-confluent mucosal breaks ≥5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential. Cumulative data collected between Day 0 and 24 and reported for time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 82 | 81
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 82 | 81
  Day 1 | 18.3 | 22.2
  Day 2: number analyzed (Participants) | 82 | 81
  Day 2 | NA — Data was not collected at this time point. | 23.5
  Day 3: number analyzed (Participants) | 82 | 81
  Day 3 | 19.5 | 24.7
  Day 4: number analyzed (Participants) | 82 | 81
  Day 4 | NA — Data was not collected at this time point. | 27.2
  Day 5: number analyzed (Participants) | 82 | 81
  Day 5 | 23.2 | 29.7
  Day 6: number analyzed (Participants) | 82 | 81
  Day 6 | 24.4 | 32.3
  Day 7: number analyzed (Participants) | 82 | 81
  Day 7 | 26.8 | 36.0
  Day 8: number analyzed (Participants) | 82 | 81
  Day 8 | 28.0 | 37.3
  Day 9: number analyzed (Participants) | 82 | 81
  Day 9 | 29.3 | 41.0
  Day 11: number analyzed (Participants) | 82 | 81
  Day 11 | 34.1 | 43.5
  Day 12: number analyzed (Participants) | 82 | 81
  Day 12 | 36.6 | 47.3
  Day 13: number analyzed (Participants) | 82 | 81
  Day 13 | NA — Data was not collected at this time point. | 51.1
  Day 14: number analyzed (Participants) | 82 | 81
  Day 14 | NA — Data was not collected at this time point. | 54.8
  Day 15: number analyzed (Participants) | 82 | 81
  Day 15 | NA — Data was not collected at this time point. | 57.3
  Day 16: number analyzed (Participants) | 82 | 81
  Day 16 | 39.0 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 82 | 81
  Day 17 | 40.2 | 58.6
  Day 18: number analyzed (Participants) | 82 | 81
  Day 18 | 43.9 | 61.1
  Day 19: number analyzed (Participants) | 82 | 81
  Day 19 | 46.3 | 63.6
  Day 20: number analyzed (Participants) | 82 | 81
  Day 20 | 47.7 | 66.3
  Day 21: number analyzed (Participants) | 82 | 81
  Day 21 | 49.1 | 67.7
  Day 22: number analyzed (Participants) | 82 | 81
  Day 22 | 52.1 | 73.4
  Day 23: number analyzed (Participants) | 82 | 81
  Day 23 | NA — Data was not collected at this time point. | 78.7
  Day 24: number analyzed (Participants) | 82 | 81
  Day 24 | NA — Data was not collected at this time point. | 89.4
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0059, Log Rank

12. Secondary Outcome: Cumulative Rate of Improvement in Heartburn in Subgroup Stratified by Endoscopic Findings (the Modified LA Classification Grade M) at Baseline
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher scores indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Cumulative rate calculated in subgroup of Grade M per modified LA classification. Modified LA classification Grade N: normal mucosa; Grade M: minimal changes to mucosa; Grade A: nonconfluent mucosal breaks <5mm in length; Grade B: non-confluent mucosal breaks ≥5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential. Cumulative data collected between Day 0 and 24 and reported for time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 163 | 157
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 163 | 157
  Day 1 | 12.9 | 23.6
  Day 2: number analyzed (Participants) | 163 | 157
  Day 2 | 14.7 | 24.9
  Day 3: number analyzed (Participants) | 163 | 157
  Day 3 | NA — Data was not collected at this time point. | 25.5
  Day 4: number analyzed (Participants) | 163 | 157
  Day 4 | 16.6 | NA — Data was not collected at this time point.
  Day 5: number analyzed (Participants) | 163 | 157
  Day 5 | NA — Data was not collected at this time point. | 27.5
  Day 6: number analyzed (Participants) | 163 | 157
  Day 6 | NA — Data was not collected at this time point. | 29.4
  Day 7: number analyzed (Participants) | 163 | 157
  Day 7 | NA — Data was not collected at this time point. | 30.7
  Day 8: number analyzed (Participants) | 163 | 157
  Day 8 | 17.8 | NA — Data was not collected at this time point.
  Day 9: number analyzed (Participants) | 163 | 157
  Day 9 | 20.9 | NA — Data was not collected at this time point.
  Day 10: number analyzed (Participants) | 163 | 157
  Day 10 | NA — Data was not collected at this time point. | 32.7
  Day 11: number analyzed (Participants) | 163 | 157
  Day 11 | 21.5 | 35.9
  Day 12: number analyzed (Participants) | 163 | 157
  Day 12 | 22.7 | 37.9
  Day 13: number analyzed (Participants) | 163 | 157
  Day 13 | 25.2 | 41.2
  Day 14: number analyzed (Participants) | 163 | 157
  Day 14 | 27.6 | 42.5
  Day 15: number analyzed (Participants) | 163 | 157
  Day 15 | 28.8 | 44.4
  Day 16: number analyzed (Participants) | 163 | 157
  Day 16 | 31.9 | 45.7
  Day 17: number analyzed (Participants) | 163 | 157
  Day 17 | 34.4 | 47.0
  Day 18: number analyzed (Participants) | 163 | 157
  Day 18 | 35.6 | 51.0
  Day 19: number analyzed (Participants) | 163 | 157
  Day 19 | 36.9 | 51.6
  Day 20: number analyzed (Participants) | 163 | 157
  Day 20 | 40.3 | 55.1
  Day 21: number analyzed (Participants) | 163 | 157
  Day 21 | 42.6 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 163 | 157
  Day 22 | 47.0 | 57.1
  Day 23: number analyzed (Participants) | 163 | 157
  Day 23 | 50.8 | 59.6
  Day 24: number analyzed (Participants) | 163 | 157
  Day 24 | NA — Data was not collected at this time point. | 63.3
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0153, Log Rank

13. Secondary Outcome: Severity of Symptoms of Heartburn in Subgroup Stratified by Endoscopic Findings (the Modified LA Classification Grade N or M) at Baseline
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. The severity of heartburn was calculated in each subgroup of the endoscopic findings where Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks <5mm in length; Grade B: non-confluent mucosal breaks ≥5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
Time Frame: Up to Week 4
Population: as for outcome 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
score on a scale
  Grade N: number analyzed (Participants) | 82 | 81
  Grade N | 1.070 [0.00 to 2.82] | 0.850 [0.00 to 3.67]
  Grade M: number analyzed (Participants) | 163 | 157
  Grade M | 1.180 [0.00 to 2.54] | 1.110 [0.00 to 2.64]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Grade N of endoscopic findings; Test type: Superiority; p = 0.0757, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1800, 95% CI 2-sided [-0.4300 to 0.0200]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Grade M of endoscopic findings; Test type: Superiority; p = 0.3837, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.0700, 95% CI 2-sided [-0.2200 to 0.0900]

14. Secondary Outcome: Percentage of Days Without Symptoms of Heartburn Stratified by Subgroup of Both the Response at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N or M)
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, higher scores indicates greater severity. The percentage was calculated in each subgroup (response; Grade N and improved, response; Grade N and not improved, response; Grade M and improved, response; Grade M and not improved) according to Criteria 1 and 2. The modified LA classification Grade N indicates the participants with normal mucosa and Grade M indicates the participants with minimal changes to the mucosa.
Time Frame: Up to Week 4
Population: FAS included participants who were randomized and received at least one dose of the study drug. Number analyzed is the number of participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of days
  Criteria 1, Grade N and Improved: number analyzed (Participants) | 28 | 39
  Criteria 1, Grade N and Improved | 93.00 [41.4 to 100.0] | 92.90 [46.4 to 100.0]
  Criteria 1, Grade N and Not Improved: number analyzed (Participants) | 54 | 41
  Criteria 1, Grade N and Not Improved | 53.60 [0.0 to 92.6] | 53.60 [0.0 to 92.9]
  Criteria 1, Grade M and Improved: number analyzed (Participants) | 55 | 60
  Criteria 1, Grade M and Improved | 89.30 [56.0 to 100.0] | 96.40 [59.3 to 100.0]
  Criteria 1, Grade M and Not Improved: number analyzed (Participants) | 108 | 95
  Criteria 1, Grade M and Not Improved | 49.05 [0.0 to 92.9] | 44.40 [0.0 to 92.9]
  Criteria 2, Grade N and Improved: number analyzed (Participants) | 59 | 61
  Criteria 2, Grade N and Improved | 69.00 [3.6 to 100.0] | 79.30 [39.3 to 100.0]
  Criteria 2, Grade N and Not Improved: number analyzed (Participants) | 23 | 20
  Criteria 2, Grade N and Not Improved | 50.00 [0.0 to 83.3] | 22.95 [0.0 to 84.0]
  Criteria 2, Grade M and Improved: number analyzed (Participants) | 109 | 113
  Criteria 2, Grade M and Improved | 73.30 [3.3 to 100.0] | 82.10 [14.3 to 100.0]
  Criteria 2, Grade M and Not Improved: number analyzed (Participants) | 54 | 44
  Criteria 2, Grade M and Not Improved | 33.90 [0.0 to 78.6] | 25.00 [0.0 to 78.6]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade N and improved response; Test type: Superiority; p = 0.6631, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.000, 95% CI 2-sided [-5.000 to 3.500]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade N and not improved response; Test type: Superiority; p = 0.5627, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.200, 95% CI 2-sided [-7.100 to 13.900]
Statistical Analysis 3: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade M and improved response; Test type: Superiority; p = 0.0042, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.700, 95% CI 2-sided [0.000 to 8.000]
Statistical Analysis 4: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade M and not improved response; Test type: Superiority; p = 0.6452, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.700, 95% CI 2-sided [-9.400 to 6.400]
Statistical Analysis 5: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade N and improved response; Test type: Superiority; p = 0.0376, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 7.400, 95% CI 2-sided [0.000 to 17.800]
Statistical Analysis 6: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade N and not improved response; Test type: Superiority; p = 0.1600, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -13.000, 95% CI 2-sided [-35.700 to 3.600]
Statistical Analysis 7: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade M and improved response; Test type: Superiority; p = 0.1032, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 3.600, 95% CI 2-sided [0.000 to 10.700]
Statistical Analysis 8: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade M and not improved response; Test type: Superiority; p = 0.2613, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -3.300, 95% CI 2-sided [-14.300 to 0.200]

15. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Improved Per Criteria 1) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N)
Description: Participants recorded the presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher scores indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 1, i.e. Improved: participants experienced heartburn on less than 2 days of 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: participants experienced heartburn on 2 days or more of the 7 days prior to Week 2 [Day 8 through Day 14]. Modified LA classification Grade N: normal mucosa and Grade M: minimal changes to the mucosa. Cumulative data was collected between Day 0 and Day 22 and is reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 11, 19, 20, and 22. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 22
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 28 | 39
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 28 | 39
  Day 1 | 53.6 | 46.2
  Day 2: number analyzed (Participants) | 28 | 39
  Day 2 | NA — Data was not collected at this time point. | 48.7
  Day 3: number analyzed (Participants) | 28 | 39
  Day 3 | 57.1 | 51.3
  Day 4: number analyzed (Participants) | 28 | 39
  Day 4 | NA — Data was not collected at this time point. | 56.4
  Day 5: number analyzed (Participants) | 28 | 39
  Day 5 | 67.9 | 61.5
  Day 6: number analyzed (Participants) | 28 | 39
  Day 6 | 71.4 | 66.7
  Day 7: number analyzed (Participants) | 28 | 39
  Day 7 | 78.6 | 74.4
  Day 8: number analyzed (Participants) | 28 | 39
  Day 8 | 82.1 | 76.9
  Day 11: number analyzed (Participants) | 28 | 39
  Day 11 | NA — Data was not collected at this time point. | 79.5
  Day 19: number analyzed (Participants) | 28 | 39
  Day 19 | 85.7 | NA — Data was not collected at this time point.
  Day 20: number analyzed (Participants) | 28 | 39
  Day 20 | NA — Data was not collected at this time point. | 82.9
  Day 22: number analyzed (Participants) | 28 | 39
  Day 22 | 89.3 | 100.0
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.9970, Log Rank

16. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Not Improved Per Criteria 1) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher scores indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 1, i.e. Improved: participants experienced heartburn on less than 2 days of 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: participants experienced heartburn on 2 days or more of 7 days prior to Week 2 [Day 8 through Day 14]. Modified LA classification Grade N indicates participants with normal mucosa and Grade M indicates participants with minimal changes to mucosa). Cumulative data was collected between Day 0 and Day 22 and is reported for following time points: Days 0, 9, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21 and 22. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 54 | 41
  Day 0 | 0.0 | 0.0
  Day 9: number analyzed (Participants) | 54 | 41
  Day 9 | 1.9 | 7.3
  Day 11: number analyzed (Participants) | 54 | 41
  Day 11 | 9.3 | 9.8
  Day 12: number analyzed (Participants) | 54 | 41
  Day 12 | 13.0 | 17.1
  Day 13: number analyzed (Participants) | 54 | 41
  Day 13 | NA — Data was not collected at this time point. | 24.4
  Day 14: number analyzed (Participants) | 54 | 41
  Day 14 | NA — Data was not collected at this time point. | 31.7
  Day 15: number analyzed (Participants) | 54 | 41
  Day 15 | NA — Data was not collected at this time point. | 36.6
  Day 16: number analyzed (Participants) | 54 | 41
  Day 16 | 16.7 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 54 | 41
  Day 17 | 18.5 | 39.0
  Day 18: number analyzed (Participants) | 54 | 41
  Day 18 | 24.1 | 43.9
  Day 19: number analyzed (Participants) | 54 | 41
  Day 19 | 25.9 | 48.8
  Day 20: number analyzed (Participants) | 54 | 41
  Day 20 | 27.9 | 51.2
  Day 21: number analyzed (Participants) | 54 | 41
  Day 21 | 30.1 | 53.8
  Day 22: number analyzed (Participants) | 54 | 41
  Day 22 | 32.4 | NA — Data was not collected at this time point.
  Day 23: number analyzed (Participants) | 54 | 41
  Day 23 | NA — Data was not collected at this time point. | 63.0
  Day 24: number analyzed (Participants) | 54 | 41
  Day 24 | NA — Data was not collected at this time point. | 81.5
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0125, Log Rank

17. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Improved Per Criteria 1) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade M)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 1, i.e. Improved: participants experienced heartburn on less than 2 days of 7 days prior to Week 2 [Day 8 through Day 14]; Not improved: participants experienced heartburn on 2 days or more of 7 days prior to Week 2 [Day 8 through Day 14]. Modified LA classification Grade N indicates participants with normal mucosa and Grade M indicates participants with minimal changes to mucosa). Cumulative data collected between Day 0 and Day 22 and is reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 11, 15, 16, 17, 18, 20, 21 and 22. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 22
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 55 | 60
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 55 | 60
  Day 1 | 38.2 | 61.7
  Day 2: number analyzed (Participants) | 55 | 60
  Day 2 | 43.6 | 65.0
  Day 3: number analyzed (Participants) | 55 | 60
  Day 3 | NA — Data was not collected at this time point. | 66.7
  Day 4: number analyzed (Participants) | 55 | 60
  Day 4 | 49.1 | NA — Data was not collected at this time point.
  Day 5: number analyzed (Participants) | 55 | 60
  Day 5 | NA — Data was not collected at this time point. | 71.7
  Day 6: number analyzed (Participants) | 55 | 60
  Day 6 | NA — Data was not collected at this time point. | 76.7
  Day 7: number analyzed (Participants) | 55 | 60
  Day 7 | NA — Data was not collected at this time point. | 80.0
  Day 8: number analyzed (Participants) | 55 | 60
  Day 8 | 52.7 | NA — Data was not collected at this time point.
  Day 11: number analyzed (Participants) | 55 | 60
  Day 11 | NA — Data was not collected at this time point. | 81.7
  Day 15: number analyzed (Participants) | 55 | 60
  Day 15 | NA — Data was not collected at this time point. | 83.3
  Day 16: number analyzed (Participants) | 55 | 60
  Day 16 | 54.5 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 55 | 60
  Day 17 | 56.4 | NA — Data was not collected at this time point.
  Day 18: number analyzed (Participants) | 55 | 60
  Day 18 | NA — Data was not collected at this time point. | 86.7
  Day 20: number analyzed (Participants) | 55 | 60
  Day 20 | 60.8 | 90.5
  Day 21: number analyzed (Participants) | 55 | 60
  Day 21 | 63.0 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 55 | 60
  Day 22 | 68.3 | NA — Data was not collected at this time point.
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0004, Log Rank

18. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Not Improved Per Criteria 1) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade M)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in a daily participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response evaluated per Criteria 1, i.e. Improved: participants experienced heartburn on < 2 days of the 7 days prior to Week 2 [Day 8 to 14]; Not improved: participants experienced heartburn on >= 2 days of 7 days prior to Week 2 [Day 8 to 14]. Modified LA classification Grade N indicates participants with normal mucosa and Grade M indicates participants with minimal changes to mucosa). Cumulative data collected between Day 0 and 24 and reported for following time points: Days 0, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 108 | 95
  Day 0 | 0.0 | 0.0
  Day 9: number analyzed (Participants) | 108 | 95
  Day 9 | 4.6 | NA — Data was not collected at this time point.
  Day 10: number analyzed (Participants) | 108 | 95
  Day 10 | NA — Data was not collected at this time point. | 3.2
  Day 11: number analyzed (Participants) | 108 | 95
  Day 11 | 5.6 | 7.4
  Day 12: number analyzed (Participants) | 108 | 95
  Day 12 | 7.4 | 10.6
  Day 13: number analyzed (Participants) | 108 | 95
  Day 13 | 11.1 | 16.0
  Day 14: number analyzed (Participants) | 108 | 95
  Day 14 | 14.8 | 18.1
  Day 15: number analyzed (Participants) | 108 | 95
  Day 15 | 16.7 | 20.2
  Day 16: number analyzed (Participants) | 108 | 95
  Day 16 | 20.4 | 22.3
  Day 17: number analyzed (Participants) | 108 | 95
  Day 17 | 23.1 | 24.5
  Day 18: number analyzed (Participants) | 108 | 95
  Day 18 | 25.0 | 28.7
  Day 19: number analyzed (Participants) | 108 | 95
  Day 19 | 26.9 | 29.8
  Day 20: number analyzed (Participants) | 108 | 95
  Day 20 | 29.9 | 33.2
  Day 21: number analyzed (Participants) | 108 | 95
  Day 21 | 32.2 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 108 | 95
  Day 22 | 36.2 | 36.4
  Day 23: number analyzed (Participants) | 108 | 95
  Day 23 | 42.0 | 40.1
  Day 24: number analyzed (Participants) | 108 | 95
  Day 24 | NA — Data was not collected at this time point. | 45.6
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.7999, Log Rank

19. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Improved Per Criteria 2) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 2, i.e. Improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was lower than during run-in period; Not improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal to or larger than during run-in period. Modified LA classification Grade N: normal mucosa and Grade M: minimal changes to mucosa). Cumulative data collected between Day 0 and 22 and reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, and 22. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 22
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 59 | 61
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 59 | 61
  Day 1 | 25.4 | 29.5
  Day 2: number analyzed (Participants) | 59 | 61
  Day 2 | NA — Data was not collected at this time point. | 31.1
  Day 3: number analyzed (Participants) | 59 | 61
  Day 3 | 27.1 | 32.8
  Day 4: number analyzed (Participants) | 59 | 61
  Day 4 | NA — Data was not collected at this time point. | 36.1
  Day 5: number analyzed (Participants) | 59 | 61
  Day 5 | 28.8 | 39.3
  Day 6: number analyzed (Participants) | 59 | 61
  Day 6 | 30.5 | 42.6
  Day 7: number analyzed (Participants) | 59 | 61
  Day 7 | 33.9 | 47.5
  Day 8: number analyzed (Participants) | 59 | 61
  Day 8 | 35.6 | 49.2
  Day 9: number analyzed (Participants) | 59 | 61
  Day 9 | NA — Data was not collected at this time point. | 52.5
  Day 11: number analyzed (Participants) | 59 | 61
  Day 11 | 40.7 | 55.7
  Day 12: number analyzed (Participants) | 59 | 61
  Day 12 | 44.1 | 59.0
  Day 13: number analyzed (Participants) | 59 | 61
  Day 13 | NA — Data was not collected at this time point. | 62.3
  Day 14: number analyzed (Participants) | 59 | 61
  Day 14 | NA — Data was not collected at this time point. | 63.9
  Day 15: number analyzed (Participants) | 59 | 61
  Day 15 | NA — Data was not collected at this time point. | 67.2
  Day 16: number analyzed (Participants) | 59 | 61
  Day 16 | 47.5 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 59 | 61
  Day 17 | 49.2 | 68.9
  Day 18: number analyzed (Participants) | 59 | 61
  Day 18 | 54.2 | 72.1
  Day 19: number analyzed (Participants) | 59 | 61
  Day 19 | 55.9 | 73.8
  Day 20: number analyzed (Participants) | 59 | 61
  Day 20 | NA — Data was not collected at this time point. | 77.5
  Day 21: number analyzed (Participants) | 59 | 61
  Day 21 | NA — Data was not collected at this time point. | 79.4
  Day 22: number analyzed (Participants) | 59 | 61
  Day 22 | 58.1 | 84.5
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0059, Log Rank

20. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Not Improved Per Criteria 2) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement was calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 2, i.e. Improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was lower than during run-in period; Not improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal to or larger than during run-in period. Modified LA classification Grade N: normal mucosa and Grade M: minimal changes to mucosa. Cumulative data was collected between Day 0 and Day 24 and is reported for following time points: Days 0, 5, 9, 11, 12, 13, 14, 19, 20, 21, 22, 23, and 24. Data not collected were shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 23 | 20
  Day 0 | 0.0 | 0.0
  Day 5: number analyzed (Participants) | 23 | 20
  Day 5 | 8.7 | NA — Data was not collected at this time point.
  Day 9: number analyzed (Participants) | 23 | 20
  Day 9 | 13.0 | 5.3
  Day 11: number analyzed (Participants) | 23 | 20
  Day 11 | 17.4 | NA — Data was not collected at this time point.
  Day 12: number analyzed (Participants) | 23 | 20
  Day 12 | NA — Data was not collected at this time point. | 10.5
  Day 13: number analyzed (Participants) | 23 | 20
  Day 13 | NA — Data was not collected at this time point. | 15.8
  Day 14: number analyzed (Participants) | 23 | 20
  Day 14 | NA — Data was not collected at this time point. | 26.3
  Day 19: number analyzed (Participants) | 23 | 20
  Day 19 | 21.7 | 31.6
  Day 20: number analyzed (Participants) | 23 | 20
  Day 20 | 26.3 | NA — Data was not collected at this time point.
  Day 21: number analyzed (Participants) | 23 | 20
  Day 21 | 30.9 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 23 | 20
  Day 22 | 35.9 | 39.2
  Day 23: number analyzed (Participants) | 23 | 20
  Day 23 | NA — Data was not collected at this time point. | 59.5
  Day 24: number analyzed (Participants) | 23 | 20
  Day 24 | NA — Data was not collected at this time point. | 100.0
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.5520, Log Rank

21. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Improved Per Criteria 2) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade M)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 2, i.e. Improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was lower than during run-in period; Not improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal or larger than during run-in period. Modified LA classification Grade N: normal mucosa and Grade M: minimal changes to mucosa. Cumulative data collected between Day 0 and 24 and reported for following time points: Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 24
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 109 | 113
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 109 | 113
  Day 1 | 19.3 | 32.7
  Day 2: number analyzed (Participants) | 109 | 113
  Day 2 | 22.0 | 34.5
  Day 3: number analyzed (Participants) | 109 | 113
  Day 3 | NA — Data was not collected at this time point. | 35.4
  Day 4: number analyzed (Participants) | 109 | 113
  Day 4 | 24.8 | NA — Data was not collected at this time point.
  Day 5: number analyzed (Participants) | 109 | 113
  Day 5 | NA — Data was not collected at this time point. | 38.1
  Day 6: number analyzed (Participants) | 109 | 113
  Day 6 | NA — Data was not collected at this time point. | 40.7
  Day 7: number analyzed (Participants) | 109 | 113
  Day 7 | NA — Data was not collected at this time point. | 42.5
  Day 8: number analyzed (Participants) | 109 | 113
  Day 8 | 26.6 | NA — Data was not collected at this time point.
  Day 9: number analyzed (Participants) | 109 | 113
  Day 9 | 30.3 | NA — Data was not collected at this time point.
  Day 10: number analyzed (Participants) | 109 | 113
  Day 10 | NA — Data was not collected at this time point. | 45.2
  Day 11: number analyzed (Participants) | 109 | 113
  Day 11 | 31.2 | 49.7
  Day 12: number analyzed (Participants) | 109 | 113
  Day 12 | 33.0 | 51.5
  Day 13: number analyzed (Participants) | 109 | 113
  Day 13 | 35.8 | 55.1
  Day 15: number analyzed (Participants) | 109 | 113
  Day 15 | 36.7 | 56.0
  Day 16: number analyzed (Participants) | 109 | 113
  Day 16 | 39.4 | 57.8
  Day 17: number analyzed (Participants) | 109 | 113
  Day 17 | 43.2 | 58.7
  Day 18: number analyzed (Participants) | 109 | 113
  Day 18 | NA — Data was not collected at this time point. | 61.4
  Day 19: number analyzed (Participants) | 109 | 113
  Day 19 | 44.1 | 62.3
  Day 20: number analyzed (Participants) | 109 | 113
  Day 20 | 48.2 | 65.1
  Day 21: number analyzed (Participants) | 109 | 113
  Day 21 | 50.6 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 109 | 113
  Day 22 | 56.1 | NA — Data was not collected at this time point.
  Day 23: number analyzed (Participants) | 109 | 113
  Day 23 | NA — Data was not collected at this time point. | 69.0
  Day 24: number analyzed (Participants) | 109 | 113
  Day 24 | NA — Data was not collected at this time point. | 75.2
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0175, Log Rank

22. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Both the Response (Not Improved Per Criteria 2) at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade M)
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe: 4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Response was evaluated per Criteria 2, i.e. Improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was lower than during run-in period; Not improved: participants experienced heartburn during treatment period up to Week 2 [Day 14] was equal to or larger than during run-in period. Modified LA classification Grade N: normal mucosa and Grade M: minimal changes to mucosa). Cumulative data was collected between Day 0 and Day 23 and is reported for following time points: Days 0, 9, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, and 23. Data not collected shown as NA=Not Applicable.
Time Frame: Day 0 to Day 23
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 54 | 44
  Day 0 | 0.0 | 0.0
  Day 9: number analyzed (Participants) | 54 | 44
  Day 9 | 1.9 | NA — Data was not collected at this time point.
  Day 12: number analyzed (Participants) | 54 | 44
  Day 12 | NA — Data was not collected at this time point. | 2.4
  Day 13: number analyzed (Participants) | 54 | 44
  Day 13 | 3.7 | 4.8
  Day 14: number analyzed (Participants) | 54 | 44
  Day 14 | 11.1 | 9.5
  Day 15: number analyzed (Participants) | 54 | 44
  Day 15 | 13.0 | 14.3
  Day 16: number analyzed (Participants) | 54 | 44
  Day 16 | 16.7 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 54 | 44
  Day 17 | NA — Data was not collected at this time point. | 16.7
  Day 18: number analyzed (Participants) | 54 | 44
  Day 18 | 20.4 | 23.8
  Day 19: number analyzed (Participants) | 54 | 44
  Day 19 | 22.3 | NA — Data was not collected at this time point.
  Day 20: number analyzed (Participants) | 54 | 44
  Day 20 | 24.3 | 29.1
  Day 21: number analyzed (Participants) | 54 | 44
  Day 21 | 26.5 | NA — Data was not collected at this time point.
  Day 22: number analyzed (Participants) | 54 | 44
  Day 22 | 29.0 | 36.2
  Day 23: number analyzed (Participants) | 54 | 44
  Day 23 | 43.2 | NA — Data was not collected at this time point.
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.7505, Log Rank

23. Secondary Outcome: Severity of Symptoms of Heartburn in Subgroup Stratified by Both the Response at Week 2 and the Endoscopic Findings (the Modified LA Classification Grade N or M)
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. The mean severity of heartburn was calculated in each subgroup (response; Grade N and improved, response; Grade N and not improved, response; Grade M and improved, response; Grade M and not improved) according to criteria 1 and 2. The modified LA classification Grade N indicates the participants with normal mucosa and Grade M indicates the participants with minimal changes to the mucosa.
Time Frame: Up to Week 4
Population: as for outcome 14
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
score on a scale
  Criteria 1, Grade N and Improved: number analyzed (Participants) | 28 | 39
  Criteria 1, Grade N and Improved | 0.510 [0.00 to 1.31] | 0.430 [0.00 to 1.56]
  Criteria 1, Grade N and Not Improved: number analyzed (Participants) | 54 | 41
  Criteria 1, Grade N and Not Improved | 1.375 [0.59 to 2.82] | 1.240 [0.14 to 2.48]
  Criteria 1, Grade M and Improved: number analyzed (Participants) | 55 | 60
  Criteria 1, Grade M and Improved | 0.420 [0.00 to 1.44] | 0.280 [0.00 to 1.20]
  Criteria 1, Grade M and Not Improved: number analyzed (Participants) | 108 | 95
  Criteria 1, Grade M and Not Improved | 1.430 [0.25 to 2.54] | 1.520 [0.14 to 2.64]
  Criteria 2, Grade N and Improved: number analyzed (Participants) | 59 | 61
  Criteria 2, Grade N and Improved | 1.000 [0.00 to 2.00] | 0.640 [0.00 to 1.68]
  Criteria 2, Grade N and Not Improved: number analyzed (Participants) | 23 | 20
  Criteria 2, Grade N and Not Improved | 1.460 [0.60 to 2.82] | 1.695 [0.48 to 3.67]
  Criteria 2, Grade M and Improved: number analyzed (Participants) | 109 | 113
  Criteria 2, Grade M and Improved | 0.890 [0.00 to 2.14] | 0.710 [0.00 to 2.04]
  Criteria 2, Grade M and Not Improved: number analyzed (Participants) | 54 | 44
  Criteria 2, Grade M and Not Improved | 1.645 [0.44 to 2.54] | 1.790 [0.43 to 2.64]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade N and improved response; Test type: Superiority; p = 0.7845, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.0300, 95% CI 2-sided [-0.2300 to 0.1600]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade N and not improved response; Test type: Superiority; p = 0.4456, Wilcoxon Rank-Sum Test; Wilcoxon Rank-Sum Test = -0.1100, 95% CI 2-sided [-0.3300 to 0.1700]
Statistical Analysis 3: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade M and improved response; Test type: Superiority; p = 0.0200, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1500, 95% CI 2-sided [-0.2900 to -0.0200]
Statistical Analysis 4: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 1, Grade M and not improved response; Test type: Superiority; p = 0.4673, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.0600, 95% CI 2-sided [-0.1000 to 0.2200]
Statistical Analysis 5: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade N and improved response; Test type: Superiority; p = 0.0095, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.2900, 95% CI 2-sided [-0.5300 to -0.0700]
Statistical Analysis 6: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade N and not improved response; Test type: Superiority; p = 0.1650, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.3100, 95% CI 2-sided [-0.1600 to 0.7100]
Statistical Analysis 7: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade M and improved response; Test type: Superiority; p = 0.2475, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.0800, 95% CI 2-sided [-0.2400 to 0.0700]
Statistical Analysis 8: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for Criteria 2, Grade M and not improved; Test type: Superiority; p = 0.2367, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 0.1300, 95% CI 2-sided [-0.0900 to 0.3200]

24. Secondary Outcome: Percentage of Days Without Symptoms of Heartburn in Subgroup Stratified by Response (Improved or Not Improved) to Acid Suppressants in Participants Who Had a Medication History
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, higher score indicates greater severity. The percentage was calculated in each subgroup of the response (improved or not improved) in the participants who had a medication history of any of acid suppressants. The acid suppressants include proton pump inhibitors [PPIs], histamine H2-receptor antagonists [H2RAs], or other agents [anticholinergics or anti-gastrin drugs].
Time Frame: Up to Week 4
Population: as for outcome 14
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of days
  Improved: number analyzed (Participants) | 83 | 88
  Improved | 61.30 [0.0 to 100.0] | 71.40 [0.0 to 100.0]
  Not Improved: number analyzed (Participants) | 8 | 5
  Not Improved | 49.30 [0.0 to 100.0] | 80.80 [39.3 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for improved response; Test type: Superiority; p = 0.1885, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 5.500, 95% CI 2-sided [-2.700 to 14.300]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for not improved response; Test type: Superiority; p = 0.2337, Wilcoxon Rank-Sum Test; Wilcoxon Rank-Sum Test = 25.600, 95% CI 2-sided [-19.200 to 75.000]

25. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Improved) to Acid Suppressants in Participants Who Had a Medication History
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Cumulative improvement rate calculated in each subgroup of the response (improved or not improved) in participants who had medication history of any of acid suppressants. Acid suppressants include proton pump inhibitors [PPIs], histamine H2-receptor antagonists [H2RAs], or other agents [anticholinergics or anti-gastrin drugs]. Cumulative data collected between Day 0 and Day 23 and is reported for following time points: Days 0, 1, 2, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22 and 23. Data not collected were shown as NA=Not Applicable.
Time Frame: Up to Week 4
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 83 | 88
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 83 | 88
  Day 1 | 13.3 | 25.0
  Day 2: number analyzed (Participants) | 83 | 88
  Day 2 | 15.7 | 26.2
  Day 4: number analyzed (Participants) | 83 | 88
  Day 4 | 18.1 | NA — Data was not collected at this time point.
  Day 5: number analyzed (Participants) | 83 | 88
  Day 5 | 20.5 | NA — Data was not collected at this time point.
  Day 6: number analyzed (Participants) | 83 | 88
  Day 6 | 21.7 | 27.3
  Day 7: number analyzed (Participants) | 83 | 88
  Day 7 | NA — Data was not collected at this time point. | 28.5
  Day 8: number analyzed (Participants) | 83 | 88
  Day 8 | 22.9 | 29.6
  Day 9: number analyzed (Participants) | 83 | 88
  Day 9 | 25.3 | NA — Data was not collected at this time point.
  Day 10: number analyzed (Participants) | 83 | 88
  Day 10 | NA — Data was not collected at this time point. | 30.8
  Day 11: number analyzed (Participants) | 83 | 88
  Day 11 | NA — Data was not collected at this time point. | 35.4
  Day 12: number analyzed (Participants) | 83 | 88
  Day 12 | 26.5 | NA — Data was not collected at this time point.
  Day 13: number analyzed (Participants) | 83 | 88
  Day 13 | NA — Data was not collected at this time point. | 41.2
  Day 14: number analyzed (Participants) | 83 | 88
  Day 14 | 28.9 | 42.3
  Day 15: number analyzed (Participants) | 83 | 88
  Day 15 | 30.1 | 43.5
  Day 16: number analyzed (Participants) | 83 | 88
  Day 16 | 31.3 | NA — Data was not collected at this time point.
  Day 17: number analyzed (Participants) | 83 | 88
  Day 17 | 32.6 | NA — Data was not collected at this time point.
  Day 18: number analyzed (Participants) | 83 | 88
  Day 18 | 33.8 | 46.9
  Day 19: number analyzed (Participants) | 83 | 88
  Day 19 | 35.0 | NA — Data was not collected at this time point.
  Day 20: number analyzed (Participants) | 83 | 88
  Day 20 | 36.3 | 49.4
  Day 21: number analyzed (Participants) | 83 | 88
  Day 21 | NA — Data was not collected at this time point. | 50.8
  Day 22: number analyzed (Participants) | 83 | 88
  Day 22 | 41.6 | 54.5
  Day 23: number analyzed (Participants) | 83 | 88
  Day 23 | 48.9 | 61.0
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0811, Log Rank

26. Secondary Outcome: Cumulative Rate of Improvement in Symptoms of Heartburn in Subgroup Stratified by Response (Not Improved) to Acid Suppressants in Participants Who Had a Medication History
Description: Participants recorded presence and severity (Without symptom [No symptom:0, No hindrance to daily activities:1], With symptom [Mild:2, Moderate:3, Severe:4]) of heartburn in participant diary. Score range was 0-4, higher score indicates greater severity. Cumulative rate of improvement calculated as percentage of participants who experienced symptom improvement. Cumulative improvement rate calculated in each subgroup of the response (improved or not improved) in participants who had medication history of any of acid suppressants. Acid suppressants include proton pump inhibitors [PPIs], histamine H2-receptor antagonists [H2RAs], or other agents [anticholinergics or anti-gastrin drugs]. Cumulative data was collected between Day 0 and Day 23 and is reported for following time points: Days 0, 1, 5, 9, 16, 19, and 20. Data not collected were shown as NA=Not Applicable.
Time Frame: Up to Week 4
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
percentage of participants
  Day 0: number analyzed (Participants) | 8 | 5
  Day 0 | 0.0 | 0.0
  Day 1: number analyzed (Participants) | 8 | 5
  Day 1 | 25.0 | 40.0
  Day 5: number analyzed (Participants) | 8 | 5
  Day 5 | NA — Data was not collected at this time point. | 60.0
  Day 9: number analyzed (Participants) | 8 | 5
  Day 9 | NA — Data was not collected at this time point. | 80.0
  Day 16: number analyzed (Participants) | 8 | 5
  Day 16 | 37.5 | NA — Data was not collected at this time point.
  Day 19: number analyzed (Participants) | 8 | 5
  Day 19 | NA — Data was not collected at this time point. | 100.0
  Day 20: number analyzed (Participants) | 8 | 5
  Day 20 | 50.0 | NA — Data was not collected at this time point.
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Test type: Superiority; p = 0.0288, Log Rank

27. Secondary Outcome: Severity of Symptoms of Heartburn in Subgroup Stratified by Response (Improved or Not Improved) to Acid Suppressants in Participants Who Had a Medication History
Description: Heartburn symptoms were collected by participant diaries. Participants recorded the presence and severity (Without symptom [No symptom: 0, No hindrance to daily activities: 1], With symptom [Mild: 2, Moderate: 3, Severe: 4]) of heartburn in a daily participant diary. The score range was 0-4, with the higher scores reflecting the greater severity. The mean severity of heartburn was calculated in each subgroup of the response (improved or not improved) in the participants who had a medication history of any of acid suppressants. The acid suppressants include proton pump inhibitors [PPIs], histamine H2-receptor antagonists [H2RAs], or other agents [anticholinergics or anti-gastrin drugs].
Time Frame: Up to Week 4
Population: as for outcome 14
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | TAK-438 10 mg
Number analyzed (Participants) | 245 | 238
score on a scale
  Improved: number analyzed (Participants) | 83 | 88
  Improved | 1.150 [0.00 to 2.82] | 1.040 [0.00 to 3.67]
  Not Improved: number analyzed (Participants) | 8 | 5
  Not Improved | 1.280 [0.00 to 2.00] | 1.030 [0.18 to 1.68]
Statistical Analysis 1: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for improved response; Test type: Superiority; p = 0.1488, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -0.1700, 95% CI 2-sided [-0.4200 to 0.0400]
Statistical Analysis 2: Comparison: Placebo vs TAK-438 10 mg; Statistical analysis for not improved response; Test type: Superiority; p = 0.3778, Wilcoxon Rank-Sum Test; Wilcoxon Rank-Sum Test = -0.4400, 95% CI 2-sided [-1.5700 to 0.6900]

ADVERSE EVENTS:
Time Frame: Up to Week 4
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-438 10 mg
All-Cause Mortality (participants affected / at risk) | 0/245 | 0/238
Serious Adverse Events (participants affected / at risk) | 1/245 | 0/238
Other Adverse Events (participants affected / at risk) | 12/245 | 10/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=245) | TAK-438 10 mg (N=238)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=245) | TAK-438 10 mg (N=238)
Viral upper respiratory tract infection (Infections and infestations) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02954848/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT02954848/SAP_001.pdf